CLINICAL TRIAL: NCT06927986
Title: A Randomized, Open-label, Multi-center, Phase III Clinical Study Comparing SYS6010 With Platinum-based Chemotherapy in the Treatment of EGFR-mutated Locally Advanced or Metastatic Non-small Cell Lung Cancer After Failure of EGFR TKI Treatment
Brief Title: Phase III Trial of SYS6010 Versus Platinum-based Chemotherapy for EGFR-mutated NSCLC（SYNSTAR01）
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6010-011
Record Dates: First submitted 2025-03-12; First posted 2025-04-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: EGFR-mutated Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: SYS6010,Q3W This is a randomized, open-label, multi-center, phase III clinical study, aiming to evaluate the efficacy and safety of SYS6010 versus platinum-based chemotherapy in participants with EGFR-mutated locally advanced or metastatic NSCLC who have failed EGFR TKI therapy. Approximately 380 participants are planned to be enrolled, who will be randomly assigned in a 1:1 ratio to the experimental group: SYS6010, and the control group: pemetrexed + cisplatin/carboplatin. Randomization stratification factors include: presence of brain metastasis (yes or no), received third-generation EGFR TKI treatment before (yes or no)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6010 (Experimental)
  Interventions: Drug: SYS6010
- Platinum-containing chemotherapy (Active Comparator): Pemetrexed injection 500 mg/m^2 + cisplatin 75 mg/m^2 or carboplatin (AUC=5, Calvert formula) administered via intravenous infusion，Q3W
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: SYS6010 — SYS6010,Q3W
  Arms: SYS6010
Drug: Pemetrexed — Pemetrexed injection 500 mg/m^2 administered via intravenous infusion，Q3W
  Arms: Platinum-containing chemotherapy
Drug: Cisplatin — Cisplatin 75 mg/m^2 administered via intravenous infusion，Q3W
  Arms: Platinum-containing chemotherapy
Drug: Carboplatin — Carboplatin (AUC=5, Calvert formula) administered via intravenous infusion，Q3W
  Arms: Platinum-containing chemotherapy

SUMMARY:
To evaluate the efficacy and safety of SYS6010 versus platinum-based chemotherapy in participants with EGFR-mutated locally advanced or metastatic non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, phase III clinical study, aiming to evaluate the efficacy and safety of SYS6010 versus platinum-based chemotherapy in participants with EGFR-mutated locally advanced or metastatic NSCLC who have failed EGFR TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 (inclusive) years old, male or females;
2. Patients with pathologically confirmed locally advanced or metastatic NSCLC, including those with stage IIIB or IIIC based on 8th edition of the AJCC staging system who are not suitable for surgical resection or radical chemoradiotherapy, or those with stage IV NSCLC. Patients with EGFR-mutated locally advanced or metastatic NSCLC who have failed EGFR TKI therapy，whereas patients progressed on first- or second-generation EGFR-TKIs must have also progressed on third-generation EGFR-TKIs if T790M mutation was detected as postive status.
3. Presence of at least one EGFR-sensitive mutation;
4. At least one measurable lesion confirmed by CT or MRI scan according to RECIST v1.1 criteria;
5. ECOG performance status of 0-1;
6. Life expectancy ≥ 3 months;
7. Major organ function must meet the following criteria within 7 days prior to randomizationn (No component transfusion, G-CSF, TPO, IL-11, or EPO within 2 weeks prior to randomization):

   Hematology： Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥100×10^9/L; Hemoglobin (HGB) ≥100g/L. Renal function Cr：≤ 1.5 × upper limit of normal (ULN) and creatinine clearance ≥ 50 mL/min; Liver function Serum total bilirubin (TBIL) ：≤ 1.5 × ULN, ≤ 3 × ULN for patients with Gilbert syndrome/metastases to liver Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)：≤ 2.5 × ULN, ≤ 5 × ULN for patients with metastases to liver Coagulation function Coagulation function Activated partial thromboplastin time (APTT) and international normalised ratio (INR)： ≤1.5×ULN
8. Women of childbearing potential must have a negative blood pregnancy test within 7 days prior to randomization. Participants must agree to use effective contraception from the time of signing the informed consent form until 7 months after the last dose; during this period, women should not be breastfeeding, and men should avoid donating sperm;
9. Voluntarily participate in this clinical study, understand the study procedures, and be able to sign a written informed consent form.

Exclusion Criteria:

1. Histologically or cytologically confirmed combined small cell lung cancer,squamous cell carcinoma, neuroendocrine carcinoma,or carcinosarcoma
2. Patients with meningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, or active CNS metastasis. Patients with supratentorial and/or cerebellar metastasis (i.e., without mesencephalon, pons, or medulla involvement) who have received local treatment, have achieved stability for at least 2 weeks prior to randomization (imaging shows no new brain metastasis or enlargement of existing brain metastasis, and all neurologic symptoms have stabilized or returned to normal), and do not require corticosteroid therapy or are receiving prednisone at a daily dose of ≤10 mg or equivalent doses of other corticosteroids, can participate in the study;
3. Patients with a history of other malignant tumors within 3 years prior to randomization, except for the following conditions: cured skin basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, and cervical carcinoma in situ, etc.;
4. Patients who are known to be allergic to any component of SYS6010 or to humanized monoclonal antibody products; allergic to carboplatin, cisplatin, or pemetrexed, or have contraindications for their use;
5. AEs caused by prior anti-tumor treatment have not recovered to ≤ Grade 1 (excluding Grade 2 alopecia, peripheral neurotoxicity, and other toxicities judged by the investigator to have no safety risk) according to NCI-CTCAE v5.0;
6. Previously received systemic anti-tumor therapy for locally advanced or metastatic non-squamous NSCLC other than EGFR TKI; patients who have previously received adjuvant/neoadjuvant chemotherapy and experienced disease progression more than 12 months after the end of treatment are allowed to be included;
7. Patients who have not met the corresponding washout period requirements for the following medications or treatments should be excluded:

   1. Major surgery (excluding needle biopsy)：At least 4 weeks
   2. Small molecule targeted drugs, traditional Chinese medicines with anti-tumor indications, palliative radiation or local therapy：At least 2 weeks
   3. intravenous injection of antibiotics, antifungals, or antivirals：At least 2 weeks
   4. Investigational product and Live attenuated vaccine：At least 4 weeks
   5. Strong CYP3A4 inducers or inhibitors ,OATP1B1 and OATP1B3 inhibitors：At least 2 weeks
8. History of severe cardiovascular or cerebrovascular disease within 6 months prior to randomization, including but not limited to:

   1. Presence of severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, third-degree atrioventricular block, Fridericia-corrected QT interval > 470 ms (Fridericia formula: QTcF = QT/RR0.33, RR = 60/heart rate);
   2. History of myocardial infarction, unstable angina pectoris, aortic dissection, angioplasty, or coronary artery bypass;
   3. NYHA class II or higher cardiac failure, LVEF<50% at screening;
   4. Stroke or other Grade 3 or higher cardiovascular and cerebrovascular events;
   5. Pulmonary embolism;
9. Imaging examination suggests tumor invasion of the cervical, thoracic, and abdominal great vessels; and the investigator assessed that there was no risk of bleeding.
10. Patients who have a history of ILD/non-infectious pneumonitis treated with corticosteroids in the past, currently have ILD/non-infectious pneumonitis, for whom imaging examinations at screening cannot rule out ILD/non-infectious pneumonitis, or whose pulmonary function test indicates severe ventilatory dysfunction and/or decreased diffusion capacity;
11. Presence of severe infections within 4 weeks prior to randomization, including but not limited to bacteraemia requiring hospitalisation, severe pneumonia, active pulmonary tuberculosis infection, etc.; presence of active infections requiring systemic antibiotics within 2 weeks prior to randomization;
12. Previous permanent discontinuation of EGFR-targeted therapy due to skin toxicity, or currently have skin diseases requiring oral or intravenous medication;
13. History of ulcerative colitis or Crohn's disease;
14. Pleural effusion or pericardial effusion requiring clinical intervention within 2 weeks prior to randomization;
15. Active HBV or HCV infection (hepatitis B surface antigen and/or hepatitis B core antibody positive and HBV DNA copies ≥ 1×104 copies/mL or ≥ 2000 IU/mL, HCV antibody positive and HCV RNA above the lower limit of detection of the analytical procedure). Note: For HBsAg-positive patients, it is recommended to start antiviral therapy before randomization, nucleoside analogues are recommended, such as entecavir, tenofovir disoproxil;
16. History of immunodeficiency (including positive HIV test, other acquired or congenital immunodeficiency diseases), history of allogeneic stem cell or organ transplant;
17. Other conditions that the investigator deems unsuitable for participation in this clinical study (such as mental disorders, macular cystoid oedema, severe corneal disorders, uncontrolled or poorly controlled hypertension and diabetes mellitus).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by independent review committee (IRC) | Up to approximately 1.5 years
  Defined as the time from randomisation until the date of objective disease progression or death was assessed by IRC according to RECIST 1.1

SECONDARY OUTCOMES:
Investigator-assessed PFS | Up to approximately 1.5 years
  Defined as the time from randomisation until the date of objective disease progression or death was assessed by investigator according to RECIST 1.1
Disease Control Rate (DCR) | Up to approximately 2 years
  Defined as the percentage of subjects who have a best overall response of CR or PR or SD based on IRC and investigator according to RECIST 1.1
Objective response rate (ORR) | Up to approximately 1.5 years
  : Defined as the proportion of patients with response (including CR and PR) assessed by the investigator and the IRC according to RECIST v1.1.
Overall Survival (OS) | Up to approximately 2 years
  Defined as the time from randomization until death from any cause
Incidence of adverse events (AEs) | Up to approximately 2 years
  AEs graded by CTCAE version 5.0
Serious adverse events (SAEs) | Up to approximately 2 years
  SAEs graded by CTCAE version 5.0
EORTC QLQ-LC13 questionnaire | Up to approximately 2 years
  EORTC QLQ-LC13 incorporates one multi-item scale to assess dyspnoea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and haemoptysis.
EORTC QLQ-30 questionnaire | Up to approximately 2 years
  EORTC QLQ-C30 is designed to measure cancer patients' physical, psychological and social functions.
Plasma concentrations of toxin-bound antibodies | Up to approximately 2 years
  Tests are conducted after single and continuous administration of SYS6010.
Plasma concentrations of total antibodies | Up to approximately 2 years
  Tests are conducted after single and continuous administration of SYS6010.
Plasma concentrations of free toxin (JS-1) | Up to approximately 2 years
  Tests are conducted after single and continuous administration of SYS6010.
anti-SYS6010 antibodies (ADA) | Up to approximately 2 years
  Incidence of SYS6010 anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China